CLINICAL TRIAL: NCT00831220
Title: Endothelial Dysfunction in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Dr. Ernest Sala, Servei de Pneumologia, Hospital Universitari Son Dureta
Other Study IDs: PI04/1946
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Endothelial Dysfunction
Keywords: COPD; exacerbations; EPCs; Erythropoietin; C-RP; COPD and endothelial dysfunction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Patients with a COPD exacerbation
- 2: Patients with stable COPD
- 3: Smokers or former smokers
- 4: Never smokers

SUMMARY:
Objective: To investigate the potential role of endothelial dysfunction as a pathogenic mechanism of cardiovascular events in COPD. Hypothesis: endothelial function is abnormal in patients with COPD, particularly during exacerbations of the disease. Design: prospective and controlled study performed in an university hospital. Population: we compare 4 groups of subjects, 44 patients with stable COPD, 35 patients with acute exacerbation of COPD, 10 smokers or former smokers with normal lung function and 10 never smokers matched by physical activity and BMI. Study variables: a) clinical variables: clinical information, physical examination, pulmonary function tests, ECG and sputum culture; b) Biological variables: number of Circulating Endothelial Progenitor Cells, vascular growth factors (vascular endothelial growht factor and erythropoietin), systemic inflammation (C-reactive protein, white blood cells), peripheral venous blood test (including hemogram, biochemical analysis with glycemia, cholesterol, LDLcol, HDLcol); and c) systemic vascular reactivity assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to very severe COPD admitted in the hospital because of an exacerbation, and,
* Patients with moderate to very severe COPD in stable condition.

Exclusion Criteria:

* Patients with an exacerbation of COPD who needed invasive or non invasive mechanical ventilation
* Patients with other chronic inflammatory diseases.
* Patients with other acute or active chronic systemic disease such as heart failure, renal insufficiency, etc.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an exacerbation of COPD admitted to our hospital, stable COPD recruited in an ambulatory basis, smokers or former smokers and never smokers recruited in our laboratory.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2005-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Sala, MD, Principal Investigator — Servei de Pneumologia, Hospital Universitari Son Dureta
Locations (1):
- Hospital Universitari Son Dureta, Palma Mallorca, Balearic Islands, Spain